CLINICAL TRIAL: NCT02670252
Title: Busulfan Plus Cyclophosphamide vs Total Body Irradiation Plus Cyclophosphamide Conditioning Regimen for Standard-risk Acute Lymphocytic Leukemia Undergoing HLA-matched Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: BuCY vs TBICY Conditioning Regimen for Standard-risk ALL Undergoing Allo-HSCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Xiangya Hospital of Central South University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Second Provincial General Hospital (Other); The Affiliated Hospital of Qingdao University (Other); First People's Hospital of Chenzhou (Other); Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUCY vs TBICY-ALL-2016
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Busulfan; Total Body Irradiation; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Busulfan; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BUCY (Experimental): For standard-risk ALL undergoing HLA-matched allo-HSCT，BUCY conditioning regimen was BU 3.2 mg/kg/day on days -7 and -4；CY 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)
- TBICY (Active Comparator): For standard-risk ALL undergoing HLA-matched allo-HSCT，TBICY conditioning regimen was 4.5 Gy TBI/day on days -5 and -4；CY 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Cyclophosphamide (CY); Radiation: Total Body Irradiation (TBI)

INTERVENTIONS:
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4.
  Arms: BUCY
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.
Radiation: Total Body Irradiation (TBI) — Total Body Irradiation was given 4.5 Gy TBI/day on days -5 and -4.
  Arms: TBICY

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) appears to be an efficient tool to cure standard-risk acute lymphocytic leukemia (ALL) in first CR (CR1) but the choice between BU-based or TBI-based conditioning regimens still remains controversial. In this study, the safety and efficacy of BUCY and TBICY myeloablative conditioning regimens in patients undergoing allo-HSCT for ALL in CR1 are evaluated.

DETAILED DESCRIPTION:
Allo-HSCT appears to be an efficient tool to cure standard-risk ALL in CR1. The conditioning regimen with BUCY or TBICY is considered as the standard myeloablative regimen for ALL in CR1, but the choice between BU-based or TBI-based conditioning regimen still remains controversial.In order to analyze the impact of conditioning regimen on long-term survival and relapse, in this study, the safety and efficacy of BUCY and TBICY myeloablative conditioning regimens in patients undergoing allo-HSCT for ALL in CR1 are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Standard-risk ALL
* Achieving CR1
* Undergoing HLA-matched allo-HSCT (related or unrelated)

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 2 year

SECONDARY OUTCOMES:
leukemia relapse rate | 2 year
disease-free survival (DFS) | 2 year
transplant-related mortality (TRM) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] de Berranger E, Cousien A, Petit A, Peffault de Latour R, Galambrun C, Bertrand Y, Salmon A, Rialland F, Rohrlich PS, Vannier JP, Lutz P, Yakouben K, Duhamel A, Bruno B, Michel G, Dalle JH. Impact on long-term OS of conditioning regimen in allogeneic BMT for children with AML in first CR: TBI+CY versus BU+CY: a report from the Societe Francaise de Greffe de Moelle et de Therapie Cellulaire. Bone Marrow Transplant. 2014 Mar;49(3):382-8. doi: 10.1038/bmt.2013.185. Epub 2013 Dec 9. PMID 24317131
- [Derived] Zhang H, Fan Z, Huang F, Han L, Xu Y, Xu N, Deng L, Wang S, Lin D, Luo X, Zhang Q, Liu X, Li X, Liang X, Xie S, Qu H, Yu S, Zhou H, Shi P, Xuan L, Lin R, Liu H, Jin H, Sun J, Liu Q. Busulfan Plus Cyclophosphamide Versus Total Body Irradiation Plus Cyclophosphamide for Adults Acute B Lymphoblastic Leukemia: An Open-Label, Multicenter, Phase III Trial. J Clin Oncol. 2023 Jan 10;41(2):343-353. doi: 10.1200/JCO.22.00767. Epub 2022 Sep 9. PMID 36084276